CLINICAL TRIAL: NCT04986007
Title: Addressing Nocturnal Sleep/Wake Effects on Risk of Suicide in Older Adults (ANSWERS-OA): A Pilot, Open-Label, Randomized Controlled Trial of Digital Cognitive Behavioral Therapy for Insomnia
Brief Title: Addressing Nocturnal Sleep/Wake Effects on Risk of Suicide in Older Adults
Acronym: ANSWERS-OA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failure.
Sponsor: MICHAEL A GRANDNER (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, MICHAEL A GRANDNER, Associate Professor of Psychiatry, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANSWERS-OA
Record Dates: First submitted 2021-05-24; First posted 2021-08-02 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Sleep Initiation and Maintenance Disorders; Suicidal Ideation
Keywords: Randomized Clinical Trial; digital Cognitive Behavioral Therapy for Insomnia; Older Adults; Suicidal Ideation; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: A randomized parallel clinical trial of digital cognitive behavioral therapy for insomnia versus waitlist control with subsequent crossover to digital cognitive behavioral therapy for insomnia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital Cognitive Behavioral Therapy for Insomnia (Experimental): Following baseline evaluation, participants in this group will receive 8 weeks of digital Cognitive Behavioral Therapy for Insomnia delivered using Sleep Healthy Using the Internet (SHUTi). After the interim assessment, participants will then crossover to 8 weeks of active monitoring.
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy for Insomnia
- Waitlist Control (No Intervention): Following baseline evaluation, participants in this group will undergo weekly monitoring of insomnia and suicidal ideation for 8 weeks. Participants will continue whatever treatments they are currently receiving, but will receive no specific instructions or behavioral interventions for insomnia. After the interim assessment, participants will then crossover to receive digital Cognitive Behavioral Therapy for Insomnia.

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy for Insomnia — Digital cognitive behavioral therapy for insomnia is an automated, internet-based delivery system for the core components of cognitive behavioral therapy for insomnia (CBT-I). For this trial, dCBT-I will be delivered using Sleep Healthy Using the Internet (SHUTi), which delivers the core content of CBT-I in 6 interactive lessons called Cores: Getting Ready; Sleep Scheduling; Sleep Practices; Thinking Differently; Sleep Hygiene; and Moving On. The primary therapeutic approaches deployed through these cores are stimulus control and sleep restriction. The minimum acceptable dose for this study is completion of 4 out of 6 cores; completion of fewer than 4 cores will be considered a dropout.
  Other Names: dCBT-I; SHUTi; Sleep Health Using the Internet
  Arms: digital Cognitive Behavioral Therapy for Insomnia

SUMMARY:
Suicide is a leading cause of death in the US, and insomnia is a risk factor for suicidal thoughts and behaviors. In older adults, suicide is associated with impaired cognitive functioning, and insomnia, which is more prevalent in older adults, is also linked to disrupted cognition. However, there is limited evidence on whether treatment of insomnia can improve suicidal ideation (with or without improving cognition), and no evidence specifically in older adults. Additionally, no studies have investigated digital cognitive behavioral therapy for insomnia (dCBT-I) in this populations. Consequently, this study will help inform future study designs and provide preliminary data on whether dCBT-I is effective for suicidal thinking in older adults.

DETAILED DESCRIPTION:
The primary goal of this pilot trial is to establish the feasibility and preliminary safety of implementing dCBT-I in older adults with insomnia and suicidal ideation. Secondary goals include estimating the potential efficacy and durability of dCBT-I for insomnia and suicidal ideation in this population, as well as evaluating neurocognitive functioning as a mediator/moderator of treatment response. To accomplish this, individuals 65 and older with insomnia and recent suicidal ideation will be recruited to either 12 weeks of treatment (dCBT-I) or waitlist control (WLC). After completion of dCBT-I, individuals in WLC will crossover to dCBT-I (WLC + dCBT-I). All participants will be re-evaluated at 6- and 12-months post-treatment.

The primary aims for this project are as follows:

Aim 1: Evaluate whether dCBT-I is a feasible intervention for older adults with insomnia and suicidal ideation. This will be assessed by subject participation and adherence to dCBT-I, evaluation of technological or cognitive barriers to accessing treatment, and by recruitment and dropout outcomes.

Aim 2: Investigate whether dCBT-I is safe for older adults with suicidal ideation. This will be measured by comparing post-treatment insomnia, depression, anxiety, and cognitive outcomes and spontaneous adverse event reports between dCBT-I and WLC, as well as post-treatment responses to the Side Effect Rating Scale - Patient Self Report (SERS-Pat) form.

The secondary aims for this project are as follows:

Aim 3: Explore whether dCBT-I can reduce suicidal ideation in older adults. While the investigators anticipate that dCBT-I will reduce suicidal ideation in older adults with insomnia, gathering preliminary data for effect size estimates will allow us to appropriately power future studies. Suicidal ideation will be measured pre-/post-treatment using the Columbia Suicide Severity Rating Scale (CSSRS) as well as weekly throughout treatment using self-report ratings of suicidal ideation severity. Comparisons will be dCBT-I vs. WLC (between groups) and WLC vs. WLC + dCBT-I (within group) using linear mixed-effects or generalized estimating equations models.

Aim 4: Assess the durability of dCBT-I treatment on suicidal ideation in older adults. Based on follow-up assessments at 6- and 12-months, the investigators will assess the potential duration of sustained improvement in suicidal ideation following dCBT-I in older adults, and how this is related to concurrent sleep continuity and quality.

Aim 5: Investigate whether changes in sleep and suicidal ideation during dCBT-I are associated with changes in neurocognition. Neurocognitive functioning will be formally assessed pre- and post-treatment using the NeuroCognitive Performance Test, a web-based neuropsychological assessment. Additionally, weekly assessment of response inhibition will occur using the Color Match task implemented as part of the same system.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 55 and older
* English speaking
* Male or female
* Current insomnia (Insomnia Severity Index score ≥ 8 during the baseline period).
* Recent suicidal ideation (endorsement of Items 1 or 2 of the Columbia Suicide Severity Rating Scale - Suicidal Ideation subscale within the past month).
* All participants must consent to a release of information between the research team and their treatment provider (either their prescribing psychiatrist, their masters-level non-trainee therapist, or their doctoral-level psychologist).

Exclusion Criteria:

* Diagnosis of bipolar disorder, any psychotic disorder, or other serious mental illness deemed a contraindication for dCBT-I.
* If a subject is taking psychotropic medication(s) (e.g., antidepressants, hypnotics), they should not have changed the dose within the past 6 weeks and should agree to not change the dose during the trial.
* If a subject is not taking psychotropic medication(s), they should be medication free for at least 6 weeks and should agree to not start a new medication for the duration of the trial.
* Suspicion or evidence of untreated sleep apnea, restless legs syndrome, or other untreated sleep disorder requiring treatment by a physician.
* Uncontrolled or unstable chronic medical conditions
* Life expectancy of less than 1 year as determined by record review and intake interview.
* Cognitive impairment sufficient to impair delivery or retention of dCBT-I as indicated by the Short Blessed Test.
* Are currently or are planning to work evening/overnight shifts.
* Lack of access to internet or technology necessary to engage in digital therapy.
* Participants who have been hospitalized for a suicide attempt or severe suicidal ideation, or who endorse any intent to commit suicide in the last 3 months must receive assent/approval from their treatment provider to participate, in addition to providing a release of information for the research team to communicate with the treatment team.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Aim 1a: Evaluate whether dCBT-I is a feasible intervention for older adults with insomnia and suicidal ideation. | Up to 24 weeks.
  Sub-aim 1a: Determine participant engagement with 10 weeks of dCBT-I. Metric: Percent of subjects enrolled who complete the 10 week treatment period
Aim 1b: Evaluate whether dCBT-I is a feasible intervention for older adults with insomnia and suicidal ideation. | Up to 24 weeks.
  Sub-aim 1b: Measure participant adherence to dCBT-I treatment. Metric: Percent of subjects who complete 4 out of 6 treatment modules.
Aim 2: Investigate whether dCBT-I is safe for older adults with suicidal ideation. | Up to 24 weeks.
  Metric: The frequency of self-reported side effects as measured by the Side Effect Rating Scale - Patient Self-Report (SERS-Pat) form. The SERS-Pat assesses 11 common side effects (with options for the patient to list others) by asking about their frequency ("Not at all", "A little more than usual", "More than usual", "Much more than usual") and their perceived relationship to treatment ("Not at all related", "Possibly related", "Probably related").

SECONDARY OUTCOMES:
Aim 3: Explore whether dCBT-I can reduce suicidal ideation in older adults. | Through study completion, an average of 1 year.
  Measurement of changes in Columbia Suicide Severity Rating Scale (CSSRS) scores from baseline. The CSSRS measures the presence and severity of suicidal thoughts and behaviors over an individual's lifetime, prior 3 months, and since last visit/interview. Questions are either yes/no or roughly range from 0-5, with higher scores reflecting more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Grandner, PhD, Principal Investigator — University of Arizona
Locations (1):
- Banner Whole Health Clinic, Tucson, Arizona, United States

REFERENCES:
- [Background] Pigeon WR, Pinquart M, Conner K. Meta-analysis of sleep disturbance and suicidal thoughts and behaviors. J Clin Psychiatry. 2012 Sep;73(9):e1160-7. doi: 10.4088/JCP.11r07586. PMID 23059158
- [Background] Bernert RA, Kim JS, Iwata NG, Perlis ML. Sleep disturbances as an evidence-based suicide risk factor. Curr Psychiatry Rep. 2015 Mar;17(3):554. doi: 10.1007/s11920-015-0554-4. PMID 25698339
- [Background] Harris LM, Huang X, Linthicum KP, Bryen CP, Ribeiro JD. Sleep disturbances as risk factors for suicidal thoughts and behaviours: a meta-analysis of longitudinal studies. Sci Rep. 2020 Aug 17;10(1):13888. doi: 10.1038/s41598-020-70866-6. PMID 32807889
- [Background] Liu RT, Steele SJ, Hamilton JL, Do QBP, Furbish K, Burke TA, Martinez AP, Gerlus N. Sleep and suicide: A systematic review and meta-analysis of longitudinal studies. Clin Psychol Rev. 2020 Nov;81:101895. doi: 10.1016/j.cpr.2020.101895. Epub 2020 Aug 8. PMID 32801085
- [Background] Zuromski KL, Cero I, Witte TK. Insomnia symptoms drive changes in suicide ideation: A latent difference score model of community adults over a brief interval. J Abnorm Psychol. 2017 Aug;126(6):739-749. doi: 10.1037/abn0000282. Epub 2017 May 29. PMID 28557509
- [Background] Hedstrom AK, Hossjer O, Bellocco R, Ye W, Trolle LY, Akerstedt T. Insomnia in the context of short sleep increases suicide risk. Sleep. 2021 Apr 9;44(4):zsaa245. doi: 10.1093/sleep/zsaa245. PMID 33216134
- [Background] Wang HE, Campbell-Sills L, Kessler RC, Sun X, Heeringa SG, Nock MK, Ursano RJ, Jain S, Stein MB. Pre-deployment insomnia is associated with post-deployment post-traumatic stress disorder and suicidal ideation in US Army soldiers. Sleep. 2019 Feb 1;42(2):zsy229. doi: 10.1093/sleep/zsy229. PMID 30508139
- [Background] Rossler W, Angst J, Ajdacic-Gross V, Haker H, Berrouiguet S, Ujeyl M, Glozier N, Hengartner MP. Sleep Disturbances and Suicidality-A Longitudinal Analysis From a Representative Community Study Over 30 Years. Front Psychiatry. 2018 Jul 16;9:320. doi: 10.3389/fpsyt.2018.00320. eCollection 2018. PMID 30061849
- [Background] Ferentinos P, Porichi E, Christodoulou C, Dikeos D, Papageorgiou C, Douzenis A. Sleep disturbance as a proximal predictor of suicidal intent in recently hospitalized attempters. Sleep Med. 2016 Mar;19:1-7. doi: 10.1016/j.sleep.2015.10.021. Epub 2015 Nov 24. PMID 27198939
- [Background] Li SX, Lam SP, Yu MW, Zhang J, Wing YK. Nocturnal sleep disturbances as a predictor of suicide attempts among psychiatric outpatients: a clinical, epidemiologic, prospective study. J Clin Psychiatry. 2010 Nov;71(11):1440-6. doi: 10.4088/JCP.09m05661gry. PMID 21114949
- [Background] Lin HT, Lai CH, Perng HJ, Chung CH, Wang CC, Chen WL, Chien WC. Insomnia as an independent predictor of suicide attempts: a nationwide population-based retrospective cohort study. BMC Psychiatry. 2018 May 2;18(1):117. doi: 10.1186/s12888-018-1702-2. PMID 29716570
- [Background] Fujino Y, Mizoue T, Tokui N, Yoshimura T. Prospective cohort study of stress, life satisfaction, self-rated health, insomnia, and suicide death in Japan. Suicide Life Threat Behav. 2005 Apr;35(2):227-37. doi: 10.1521/suli.35.2.227.62876. PMID 15843339
- [Background] Perlis ML, Grandner MA, Chakravorty S, Bernert RA, Brown GK, Thase ME. Suicide and sleep: Is it a bad thing to be awake when reason sleeps? Sleep Med Rev. 2016 Oct;29:101-7. doi: 10.1016/j.smrv.2015.10.003. Epub 2015 Oct 19. PMID 26706755
- [Background] Perlis ML, Grandner MA, Brown GK, Basner M, Chakravorty S, Morales KH, Gehrman PR, Chaudhary NS, Thase ME, Dinges DF. Nocturnal Wakefulness as a Previously Unrecognized Risk Factor for Suicide. J Clin Psychiatry. 2016 Jun;77(6):e726-33. doi: 10.4088/JCP.15m10131. PMID 27337421
- [Background] Tubbs AS, Perlis ML, Basner M, Chakravorty S, Khader W, Fernandez F, Grandner MA. Relationship of Nocturnal Wakefulness to Suicide Risk Across Months and Methods of Suicide. J Clin Psychiatry. 2020 Feb 25;81(2):19m12964. doi: 10.4088/JCP.19m12964. PMID 32097547
- [Background] Tubbs AS, Fernandez FX, Perlis ML, Hale L, Branas CC, Barrett M, Chakravorty S, Khader W, Grandner MA. Suicidal ideation is associated with nighttime wakefulness in a community sample. Sleep. 2021 Jan 21;44(1):zsaa128. doi: 10.1093/sleep/zsaa128. PMID 32614967
- [Background] Tubbs AS, Harrison-Monroe P, Fernandez FX, Perlis ML, Grandner MA. When reason sleeps: attempted suicide during the circadian night. J Clin Sleep Med. 2020 Oct 15;16(10):1809-1810. doi: 10.5664/jcsm.8662. PMID 32621577
- [Background] Munch M, Knoblauch V, Blatter K, Wirz-Justice A, Cajochen C. Is homeostatic sleep regulation under low sleep pressure modified by age? Sleep. 2007 Jun;30(6):781-92. doi: 10.1093/sleep/30.6.781. PMID 17580600
- [Background] Cajochen C, Brunner DP, Krauchi K, Graw P, Wirz-Justice A. Power density in theta/alpha frequencies of the waking EEG progressively increases during sustained wakefulness. Sleep. 1995 Dec;18(10):890-4. doi: 10.1093/sleep/18.10.890. PMID 8746397
- [Background] Verweij IM, Romeijn N, Smit DJ, Piantoni G, Van Someren EJ, van der Werf YD. Sleep deprivation leads to a loss of functional connectivity in frontal brain regions. BMC Neurosci. 2014 Jul 19;15:88. doi: 10.1186/1471-2202-15-88. PMID 25038817
- [Background] Valdez P, Ramirez C, Garcia A, Talamantes J, Cortez J. Circadian and homeostatic variation in sustained attention. Chronobiol Int. 2010 Jan;27(2):393-416. doi: 10.3109/07420521003765861. PMID 20370477
- [Background] Drummond SP, Paulus MP, Tapert SF. Effects of two nights sleep deprivation and two nights recovery sleep on response inhibition. J Sleep Res. 2006 Sep;15(3):261-5. doi: 10.1111/j.1365-2869.2006.00535.x. PMID 16911028
- [Background] Frey S, Birchler-Pedross A, Hofstetter M, Brunner P, Gotz T, Munch M, Blatter K, Knoblauch V, Wirz-Justice A, Cajochen C. Young women with major depression live on higher homeostatic sleep pressure than healthy controls. Chronobiol Int. 2012 Apr;29(3):278-94. doi: 10.3109/07420528.2012.656163. PMID 22390241
- [Background] Birchler-Pedross A, Frey S, Chellappa SL, Gotz T, Brunner P, Knoblauch V, Wirz-Justice A, Cajochen C. Higher frontal EEG synchronization in young women with major depression: a marker for increased homeostatic sleep pressure? Sleep. 2011 Dec 1;34(12):1699-706. doi: 10.5665/sleep.1440. PMID 22131608
- [Background] Niggemyer KA, Begley A, Monk T, Buysse DJ. Circadian and homeostatic modulation of sleep in older adults during a 90-minute day study. Sleep. 2004 Dec 15;27(8):1535-41. doi: 10.1093/sleep/27.8.1535. PMID 15683145
- [Background] Schmidt C, Collette F, Cajochen C, Peigneux P. A time to think: circadian rhythms in human cognition. Cogn Neuropsychol. 2007 Oct;24(7):755-89. doi: 10.1080/02643290701754158. PMID 18066734
- [Background] Wyatt JK, Ritz-De Cecco A, Czeisler CA, Dijk DJ. Circadian temperature and melatonin rhythms, sleep, and neurobehavioral function in humans living on a 20-h day. Am J Physiol. 1999 Oct;277(4 Pt 2):R1152-63. doi: 10.1152/ajpregu.1999.277.4.r1152. PMID 10516257
- [Background] May CP. Synchrony effects in cognition: the costs and a benefit. Psychon Bull Rev. 1999 Mar;6(1):142-7. doi: 10.3758/bf03210822. PMID 12199309
- [Background] Wright KP, Lowry CA, Lebourgeois MK. Circadian and wakefulness-sleep modulation of cognition in humans. Front Mol Neurosci. 2012 Apr 18;5:50. doi: 10.3389/fnmol.2012.00050. eCollection 2012. PMID 22529774
- [Background] May CP, Hasher L. Synchrony effects in inhibitory control over thought and action. J Exp Psychol Hum Percept Perform. 1998 Apr;24(2):363-79. doi: 10.1037//0096-1523.24.2.363. PMID 9554091
- [Background] Monk TH, Buysse DJ, Reynolds CF 3rd, Berga SL, Jarrett DB, Begley AE, Kupfer DJ. Circadian rhythms in human performance and mood under constant conditions. J Sleep Res. 1997 Mar;6(1):9-18. doi: 10.1046/j.1365-2869.1997.00023.x. PMID 9125694
- [Background] Boivin DB, Czeisler CA, Dijk DJ, Duffy JF, Folkard S, Minors DS, Totterdell P, Waterhouse JM. Complex interaction of the sleep-wake cycle and circadian phase modulates mood in healthy subjects. Arch Gen Psychiatry. 1997 Feb;54(2):145-52. doi: 10.1001/archpsyc.1997.01830140055010. PMID 9040282
- [Background] Murray G, Allen NB, Trinder J. Mood and the circadian system: investigation of a circadian component in positive affect. Chronobiol Int. 2002 Nov;19(6):1151-69. doi: 10.1081/cbi-120015956. PMID 12511032
- [Background] Monk TH, Buysse DJ, Reynolds CF 3rd, Jarrett DB, Kupfer DJ. Rhythmic vs homeostatic influences on mood, activation, and performance in young and old men. J Gerontol. 1992 Jul;47(4):P221-7. doi: 10.1093/geronj/47.4.p221. PMID 1624698
- [Background] Brewster GS, Riegel B, Gehrman PR. Insomnia in the Older Adult. Sleep Med Clin. 2018 Mar;13(1):13-19. doi: 10.1016/j.jsmc.2017.09.002. Epub 2017 Nov 22. PMID 29412980
- [Background] Patel D, Steinberg J, Patel P. Insomnia in the Elderly: A Review. J Clin Sleep Med. 2018 Jun 15;14(6):1017-1024. doi: 10.5664/jcsm.7172. PMID 29852897
- [Background] Kay DB, Dombrovski AY, Buysse DJ, Reynolds CF, Begley A, Szanto K. Insomnia is associated with suicide attempt in middle-aged and older adults with depression. Int Psychogeriatr. 2016 Apr;28(4):613-9. doi: 10.1017/S104161021500174X. Epub 2015 Nov 10. PMID 26552935
- [Background] Richard-Devantoy S, Szanto K, Butters MA, Kalkus J, Dombrovski AY. Cognitive inhibition in older high-lethality suicide attempters. Int J Geriatr Psychiatry. 2015 Mar;30(3):274-83. doi: 10.1002/gps.4138. Epub 2014 May 12. PMID 24816626
- [Background] McGirr A, Dombrovski AY, Butters MA, Clark L, Szanto K. Deterministic learning and attempted suicide among older depressed individuals: cognitive assessment using the Wisconsin Card Sorting Task. J Psychiatr Res. 2012 Feb;46(2):226-32. doi: 10.1016/j.jpsychires.2011.10.001. Epub 2011 Oct 22. PMID 22024486
- [Background] Clark L, Dombrovski AY, Siegle GJ, Butters MA, Shollenberger CL, Sahakian BJ, Szanto K. Impairment in risk-sensitive decision-making in older suicide attempters with depression. Psychol Aging. 2011 Jun;26(2):321-330. doi: 10.1037/a0021646. PMID 21443349
- [Background] Dombrovski AY, Clark L, Siegle GJ, Butters MA, Ichikawa N, Sahakian BJ, Szanto K. Reward/Punishment reversal learning in older suicide attempters. Am J Psychiatry. 2010 Jun;167(6):699-707. doi: 10.1176/appi.ajp.2009.09030407. Epub 2010 Mar 15. PMID 20231320
- [Background] Gibbs LM, Dombrovski AY, Morse J, Siegle GJ, Houck PR, Szanto K. When the solution is part of the problem: problem solving in elderly suicide attempters. Int J Geriatr Psychiatry. 2009 Dec;24(12):1396-404. doi: 10.1002/gps.2276. PMID 19405045
- [Background] Dombrovski AY, Butters MA, Reynolds CF 3rd, Houck PR, Clark L, Mazumdar S, Szanto K. Cognitive performance in suicidal depressed elderly: preliminary report. Am J Geriatr Psychiatry. 2008 Feb;16(2):109-15. doi: 10.1097/JGP.0b013e3180f6338d. PMID 18239196
- [Background] McCall WV, Benca RM, Rosenquist PB, Youssef NA, McCloud L, Newman JC, Case D, Rumble ME, Szabo ST, Phillips M, Krystal AD. Reducing Suicidal Ideation Through Insomnia Treatment (REST-IT): A Randomized Clinical Trial. Am J Psychiatry. 2019 Nov 1;176(11):957-965. doi: 10.1176/appi.ajp.2019.19030267. Epub 2019 Sep 20. PMID 31537089
- [Background] Margolis SA, Kelly DA, Daiello LA, Davis J, Tremont G, Pillemer S, Denby C, Ott BR. Anticholinergic/Sedative Drug Burden and Subjective Cognitive Decline in Older Adults at Risk of Alzheimer's Disease. J Gerontol A Biol Sci Med Sci. 2021 May 22;76(6):1037-1043. doi: 10.1093/gerona/glaa222. PMID 32886748
- [Background] Puustinen J, Lahteenmaki R, Polo-Kantola P, Salo P, Vahlberg T, Lyles A, Neuvonen PJ, Partinen M, Raiha I, Kivela SL. Effect of withdrawal from long-term use of temazepam, zopiclone or zolpidem as hypnotic agents on cognition in older adults. Eur J Clin Pharmacol. 2014 Mar;70(3):319-29. doi: 10.1007/s00228-013-1613-6. Epub 2013 Dec 12. PMID 24337417
- [Background] Morgenthaler T, Kramer M, Alessi C, Friedman L, Boehlecke B, Brown T, Coleman J, Kapur V, Lee-Chiong T, Owens J, Pancer J, Swick T; American Academy of Sleep Medicine. Practice parameters for the psychological and behavioral treatment of insomnia: an update. An american academy of sleep medicine report. Sleep. 2006 Nov;29(11):1415-9. PMID 17162987
- [Background] Trockel M, Karlin BE, Taylor CB, Brown GK, Manber R. Effects of cognitive behavioral therapy for insomnia on suicidal ideation in veterans. Sleep. 2015 Feb 1;38(2):259-65. doi: 10.5665/sleep.4410. PMID 25515115
- [Background] Pigeon WR, Funderburk JS, Cross W, Bishop TM, Crean HF. Brief CBT for insomnia delivered in primary care to patients endorsing suicidal ideation: a proof-of-concept randomized clinical trial. Transl Behav Med. 2019 Nov 25;9(6):1169-1177. doi: 10.1093/tbm/ibz108. PMID 31271210
- [Background] Hedegaard H, Curtin SC, Warner M. Suicide Mortality in the United States, 1999-2017. NCHS Data Brief. 2018 Nov;(330):1-8. PMID 30500324
- [Background] Manber R, Simpson NS, Bootzin RR. A step towards stepped care: delivery of CBT-I with reduced clinician time. Sleep Med Rev. 2015 Feb;19:3-5. doi: 10.1016/j.smrv.2014.09.003. Epub 2014 Oct 8. No abstract available. PMID 25454675
- [Background] Christensen H, Batterham PJ, Gosling JA, Ritterband LM, Griffiths KM, Thorndike FP, Glozier N, O'Dea B, Hickie IB, Mackinnon AJ. Effectiveness of an online insomnia program (SHUTi) for prevention of depressive episodes (the GoodNight Study): a randomised controlled trial. Lancet Psychiatry. 2016 Apr;3(4):333-41. doi: 10.1016/S2215-0366(15)00536-2. Epub 2016 Jan 28. PMID 26827250
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Cheng P, Luik AI, Fellman-Couture C, Peterson E, Joseph CLM, Tallent G, Tran KM, Ahmedani BK, Roehrs T, Roth T, Drake CL. Efficacy of digital CBT for insomnia to reduce depression across demographic groups: a randomized trial. Psychol Med. 2019 Feb;49(3):491-500. doi: 10.1017/S0033291718001113. Epub 2018 May 24. PMID 29792241
- [Background] Klingman KJ, Jungquist CR, Perlis ML. Questionnaires that screen for multiple sleep disorders. Sleep Med Rev. 2017 Apr;32:37-44. doi: 10.1016/j.smrv.2016.02.004. Epub 2016 Feb 27. PMID 27013458
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Lewinsohn PM, Seeley JR, Roberts RE, Allen NB. Center for Epidemiologic Studies Depression Scale (CES-D) as a screening instrument for depression among community-residing older adults. Psychol Aging. 1997 Jun;12(2):277-87. doi: 10.1037//0882-7974.12.2.277. PMID 9189988
- [Background] Radloff LS. The use of the Center for Epidemiologic Studies Depression Scale in adolescents and young adults. J Youth Adolesc. 1991 Apr;20(2):149-66. doi: 10.1007/BF01537606. PMID 24265004
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Grandner MA, Olivier K, Gallagher R, Hale L, Barrett M, Branas C, Killgore WDS, Parthasarathy S, Gehrels JA, Alfonso-Miller P. Quantifying impact of real-world barriers to sleep: The Brief Index of Sleep Control (BRISC). Sleep Health. 2020 Oct;6(5):587-593. doi: 10.1016/j.sleh.2020.01.013. Epub 2020 May 29. PMID 32482573
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Kleiman EM, Turner BJ, Fedor S, Beale EE, Huffman JC, Nock MK. Examination of real-time fluctuations in suicidal ideation and its risk factors: Results from two ecological momentary assessment studies. J Abnorm Psychol. 2017 Aug;126(6):726-738. doi: 10.1037/abn0000273. Epub 2017 May 8. PMID 28481571
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064
- [Background] Morrison GE, Simone CM, Ng NF, Hardy JL. Reliability and validity of the NeuroCognitive Performance Test, a web-based neuropsychological assessment. Front Psychol. 2015 Nov 3;6:1652. doi: 10.3389/fpsyg.2015.01652. eCollection 2015. PMID 26579035
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Dawson DA, Grant BF, Stinson FS. The AUDIT-C: screening for alcohol use disorders and risk drinking in the presence of other psychiatric disorders. Compr Psychiatry. 2005 Nov-Dec;46(6):405-16. doi: 10.1016/j.comppsych.2005.01.006. PMID 16275207